CLINICAL TRIAL: NCT04332185
Title: Vestibular Socket Therapy With Immediate Implant Placement for Managing Compromised Fresh Extraction Sockets: A Prospective Single Arm Clinical Trial
Brief Title: Vestibular Socket Therapy in Compromised Sockets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Iman Abd-ElWahab Radi, PhD, Professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0010556
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Implant Site Reaction
Keywords: Vestibular socket therapy; bone grafting; immediate implant placement; socket preservation; bone shielding; cortical bone shield

STUDY DESIGN:
Intervention Model Description: (VST) included the following steps. a-traumatic tooth extractio. One-cm long vestibular access incision was made 3-4 mm apical to the mucogingival junction at the related socket. A subperiosteal tunnel was created connecting the socket orifice and the vestibular access incision using periotomes and micro periosteal elevators . implant was placed. A flexible cortical membrane shield that is made of cortical bone of heterologous origin of 0.6 mm thickness was introduced from the vestibular access incision reaching 1 mm below the socket orifice through the tunnel then stabilized using a micro screw to the alveolar bone. The socket gap between the implant and the shield was then packed thoroughly with particulate bone graft. A chairside-fabricated anatomical healing abutment was used to seal the socket orifice . restorative phase then took place 45 days post-surgery till the final restoration finally cemented at 2 months post-surgery and followed up for 1 and 2 years using CBCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vestibulart socket therapy (Experimental): (VST) included the following steps. a-traumatic tooth extraction, the socket curetted and rinsed with normal saline thoroughly . One-cm long vestibular access incision was made using a 15c blade 3-4 mm apical to the mucogingival junction at the related socket. A subperiosteal tunnel was created connecting the socket orifice and the vestibular access incision using periotomes and micro periosteal elevators A flexible cortical membrane shield that is made of cortical bone of heterologous origin of 0.6 mm thickness was hydrated and then trimmed and introduced from the vestibular access incision reaching 1 mm below the socket orifice through the tunnel then stabilized using a micro screw to the alveolar bone apical to the base of the socket .
  Interventions: Procedure: vestibular socket therapy

INTERVENTIONS:
Procedure: vestibular socket therapy — (VST) included the following steps. a-traumatic tooth extraction, the socket curetted and rinsed with normal saline thoroughly . One-cm long vestibular access incision was made using a 15c blade 3-4 mm apical to the mucogingival junction at the related socket. A subperiosteal tunnel was created connecting the socket orifice and the vestibular access incision using periotomes and micro periosteal elevators A flexible cortical membrane shield that is made of cortical bone of heterologous origin of 0.6 mm thickness was hydrated and then trimmed and introduced from the vestibular access incision reaching 1 mm below the socket orifice through the tunnel then stabilized using a micro screw to the alveolar bone apical to the base of the socket .

SUMMARY:
Twenty compromised post-extraction sockets were managed by VST and IMP. After tooth extraction and IMP, a vestibular incision was cut and a cortical bone shield was stabilized. The jumping gap was then filled with particulate bone graft, which was protected by a healing abutment. After 2 years labial plate thickness was evaluated at 3 levels (crestal, middle and apical) using cone beam computed tomography (CBCT). Pink esthetic core (PES), and probing depth (PD) were also measured. 2 year following implant placement, the mean differences (µ) and standard deviations (SD) were calculated. Paired t-test was used for detecting significant results at P≤.05.

DETAILED DESCRIPTION:
In this protocol, atraumatic tooth extraction was carried out using periotomes (Stoma, Storz am Mark GmbH, Emmingen-Liptingen Germany) under local anaesthesia (ARTINIBSA 4% 1:100.000. Inibsa Dental S.L.U. Barcelona, SPAIN). After that, the socket was thoroughly curetted and debrided and repeatedly irrigated with 100 ml of anti-anaerobic infusion solution of 500 mg Metronidazole (Minapharm pharmaceuticals, Egypt). The root was then trimmed to half-length, its surface cleansed with an ultrasonic cleaner , and reinserted into the socket with its crown bonded to adjacent teeth . After six days, the root was removed and VST protocol was implemented.

Vestibular socket therapy (VST) included the following steps. a-traumatic tooth extraction, the socket curetted and rinsed with normal saline thoroughly (Figure 2 a,b). One-cm long vestibular access incision was made using a 15c blade (Stoma, Storz am Mark GmbH, Emmingen-Liptingen Germany) 3-4 mm apical to the mucogingival junction at the related socket (. A subperiosteal tunnel was created connecting the socket orifice and the vestibular access incision using periotomes and micro periosteal elevators (Stoma, Storz am Mark GmbH, Emmingen-Liptingen Germany) . A prefabricated CAD CAM surgical guide was used to deliver the implant fixture (Biohorizons, Birmingham, Al, USA) to its pre-planned location 3-4 mm apical to socket base with adequate primary stability achieved using a torque wrench reaching 30 Ncm torque (Figure 2 g). A flexible cortical membrane shield that is made of cortical bone of heterologous origin of 0.6 mm thickness (OsteoBiol® Lamina , Tecnoss®, Torino, Italy) was hydrated and then trimmed and introduced from the vestibular access incision reaching 1 mm below the socket orifice through the tunnel then stabilized using a membrane tack or a micro screw to the alveolar bone apical to the base of the socket (AutoTac System Kit, Biohorizons Implant Systems, Birmingham , Alabama Inc, USA) . The socket gap between the implant and the shield was then packed thoroughly with particulate bone graft (75% autogenous bone chips and 25% deproteinized bovine bone mineral (DBBM) of equine origin, fully enzyme deantigenised (Bio-Gen Mix, Bioteck, Vicenza -Italy).

For patients exhibiting thin soft tissue phenotype (assessed using the probe transparency method) a subepithelial connective tissue graft was harvested using a single incision technique (Hürzeler MB & Weng D 1999) from the palate which and secured to the inner surface of the soft tissue tunnel wall with sutures. Finally, the vestibular incision was secured with 6/0 nylon sutures (Stoma, Storz am Mark GmbH, Emmingen-Liptingen Germany) . A chairside-fabricated anatomical healing abutment was used to seal the socket orifice . restorative phase then took place 45 days post-surgery till the final restoration finally cemented at 2 months post-surgery and followed up for 2 years using CBCT.

ELIGIBILITY:
Inclusion Criteria:

* unrestorable maxillary anterior teeth
* with adequate palatal and apical bone that allows achieving adequate implant primary stability
* compromised sockets

Exclusion Criteria:

* infection
* smokers
* systemic condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
bone thickness | 2 years
  continuous outcome

SECONDARY OUTCOMES:
Bone height | 2 years
  continuous outcome
pocket depth | 1.5 year
  continuous outcome
PES | 1.5 year
  ordinal outcome

CONTACTS AND LOCATIONS:
Overall Officials: AbdelSalam T ElAskary, Dr, BDS, Study Director — Private Practice
Locations (1):
- ElAskary and Associates Private clinic, Alexandria, Egypt